CLINICAL TRIAL: NCT05266313
Title: Contributions of a Paramedical Approach in the Prevention and Treatment of Side Effects Associated With Radical Prostatectomy (RP): "Vitality", an Onco-sexology Program
Brief Title: Contributions of a Paramedical Approach in the Prevention and Treatment of Side Effects Associated With Radical Prostatectomy
Acronym: VITALITE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21_RIPH2-06
Record Dates: First submitted 2022-02-21; First posted 2022-03-04 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Prostatic Neoplasms
Keywords: Prostatic Neoplasms; Oncosexology; Paramedics; Sexual rehabilitation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oncosexology program (Experimental): Several workshops before and after the radical prostatectomy
  Interventions: Behavioral: Oncosexology program
- Usual care (No Intervention): Usual care of the urology department for patients with prostate cancer

INTERVENTIONS:
Behavioral: Oncosexology program — Thematic workshops throughout the year
  Arms: Oncosexology program

SUMMARY:
The paramedic urology team at Martinique University Hospital has developed a "personalized rehabilitation oncosexology program for patients undergoing radical prostatectomy (RP) for localized prostate cancer". The aim of this project is to assess the effectiveness of this program by comparing the sexual quality of life 1 year after surgery between patients participating and those who do not.

DETAILED DESCRIPTION:
80% of patients undergoing radical prostatectomy report urinary incontinence and erectile dysfunction [Johanssen et al. 2011. Scandinavian Prostate Cancer Group Study]. In the West Indies, the incidence of prostate cancer is one of the highest in the world (World-standardized incidence in Martinique is 164.5 versus 88.8 per 100,000 person-years in Metropolitan France). Over 2007-2014 an average 530 new cases of prostate cancer were diagnosed each year in Martinique, representing 55% of all male cancers [Regional estimates report Public Health France, January 2018]. The prostate is a symbol of male vulnerability [French Association of Urology-Global Market Research and Public Opinion Specialist, 2006]. For other authors, virility is above all a cultural representation, and the "crisis of virility", a recomposition of male identity. Surgery on a sexual organ can alter body image and masculinity. According to Colson et al., patients treated for prostate cancer and their partners clearly place sex in first place in the importance of quality of life domains.

ELIGIBILITY:
Inclusion Criteria:

* Men diagnosed with localized prostate cancer and consulting in the urology department of Mangot Vulcin site of the Martinique University Hospital
* Patients newly diagnosed for prostate cancer and who will benefit from radical prostatectomy (regardless the technique : laparotomy, laparoscopy or robot-assisted micro-invasive surgery)
* Fluent in French or Creole
* Patients who give consent
* Patients affiliated to social security

Exclusion Criteria:

* Patients diagnosed with another tumor
* Person under legal protection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2025-03-26 (Estimated); Study Completion 2025-03-26 (Estimated)

PRIMARY OUTCOMES:
Evaluation of sexual Quality of Life: Questionnaire | Before the radical prostatectomy
  Administration of sexual of life questionnaire (SEAR for self-esteem and couple relationship)
Evaluation of sexual function: Questionnaire | Before the radical prostatectomy
  Administration of sexual function questionnaire (IIEF-type validated questionnaires)
Evaluation of sexual Quality of Life: Questionnaire | 1 Month after the radical prostatectomy
  Administration of sexual of life questionnaire (SEAR for self-esteem and couple relationship)
Evaluation of sexual function: Questionnaire | 1 Month after the radical prostatectomy
  Administration of sexual function questionnaire (IIEF-type validated questionnaires)
Evaluation of sexual Quality of Life: Questionnaire | 12 months after the radical prostatectomy
  Administration of sexual of life questionnaire (SEAR for self-esteem and couple relationship)
Evaluation of sexual function: Questionnaire | 12 months after the radical prostatectomy
  Administration of sexual function questionnaire (IIEF-type validated questionnaires)

SECONDARY OUTCOMES:
Evaluation of quality of life in its multidimensional aspect | Before the radical prostatectomy
  Administration of quality of life questionnaire (EORTC QLC C30 questionnaires)
Evaluation of quality of life for localized forms of prostate cancer | Before the radical prostatectomy
  Administration of QLQ-PR25 questionnaire (specific module intended for localized forms of prostate cancer. It is complementary to QLQ-C30 and better suited to measure the side effects of treatment.)
Evaluation of quality of life in its multidimensional aspect | 12 Month after the radical prostatectomy
  Administration of quality of life questionnaire (EORTC QLC C30 questionnaires)
Evaluation of quality of life for localized forms of prostate cancer | 12 Month after the radical prostatectomy
  Administration of QLQ-PR25 questionnaire ((specific module intended for localized forms of prostate cancer. It is complementary to QLQ-C30 and better suited to measure the side effects of treatment.)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No